CLINICAL TRIAL: NCT04870775
Title: Effectiveness of a Mindfulness Training Program for Hospital Workers During the Pandemic: A Randomised Controlled Trial
Brief Title: Effectiveness of a Mindfulness Training Program for Hospital Workers During the Pandemic.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Granada (Other)
Responsible Party: Principal Investigator, Jose A. Puertas-Gonzalez, Predoctoral Researcher, Universidad de Granada
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GESTASTRESS-Covid
Record Dates: First submitted 2021-04-29; First posted 2021-05-03 (Actual); Last update posted 2021-12-08 (Actual); Status verified 2021-12

CONDITIONS: Psychopathology
Keywords: Psychopathology; Covid-19; Mindfulness; Hospital workers
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): The intervention administered to the experimental group will be a mindfulness training program
  Interventions: Behavioral: Mindfulness Training Program
- Control group (No Intervention): The control group will not receive any intervention

INTERVENTIONS:
Behavioral: Mindfulness Training Program — Mindfulness training program to reduce psychotropathological symptoms in hospital workers
  Arms: Experimental group

SUMMARY:
The aim of this study is to reduce the negative psychological impact of the pandemic on hospital workers through mindfulness training.

DETAILED DESCRIPTION:
In the face of the recent health crisis, one group vulnerable to psychological consequences has been the hospital workers who have worked on the front line during the COVID-19 pandemic.

It is expected that subjects participating in Mindfulness training will decrease their psychopathological symptoms more than the control group.

The programa will be held in 8 sessions (1 per week) as follows:

SESSION 1:

Welcome Brief opening practice with anchoring or focus options. Presentation of mindfulness, what it is and what it is not, definition and available scientific evidence.

Guided reflection on what brought the people here. Introduction of participants and teacher. Standing yoga postures. Raisin meditation. Body scan practice Presentation of home practice Brief closing practice

SESSION 2:

Brief opening practice. Standing yoga postures. Body scanner practice Dialogue on the practices, in small groups first and then in the large group. Exercise of the 9 points: conditioning and creative response. Attentional photo sitting meditation. Presentation of the home practice Brief closing practice

SESSION 3:

Brief opening practice Meditation with attention to an attentional focus. Yoga postures on the floor Dialogue in small groups and then in the common room about the experience of the practices.

Review of the calendar of pleasant events, paying attention to how it has registered in the form of bodily sensations, thoughts and emotions.

Presentation of the home practice Brief closing practice

SESSION 4:

Brief opening practice Standing yoga postures Sitting meditation with attention to the unwanted, offering the option to pendulum, from unpleasantness to attentional focus.

Dialogue in small groups and then in the common room about the experience of the practices.

Review of the calendar of unpleasant events and connect the unpleasant experience with stress.

Brief explanation of stress physiology and reactivity. Presentation of home practice Brief closing practice

SESSION 5:

Brief opening practice. Standing yoga postures. Complete meditation alternating different focuses of attention to end with open awareness.

Dialogue in small groups and then in the common room about the experience of the practices, reflection on being in the middle of the course (achievements, expectations, challenges...).

Introduce mindfulness in any of the phases of the habit loop and in moments of reactivity. Concept of mindful pause.

Presentation of home practice Brief closing practice

SESSION 6:

Brief opening practice. Standing yoga postures. Full seated meditation, with more silence and less guidance. Dialogue in small groups and then in the common room about the experience of the practices, introducing reflections on engagement with the practice and its effects and challenges.

Guided reflection on a difficult communication situation and interactive dialogue from there.

Presentation of home practice Brief closing practice

SESSION 7:

Brief opening practice. Movement practice: encouraging simplicity and exploration of boundaries. Participants are invited to guide some of them.

Sitting meditation, with more silence and less guidance. Dialogue in small groups and then in the common room about the experience of the day's practice.

Reflection on how people relate to their environment and the choices people make around technology, social networking, media and what effects those choices have.

Presentation of home practice Brief closing practice

SESSION 8:

Brief opening practice. Body scanning practice Small group discussion and then in the common room about the home practice. Writing a letter to the "future self" after reflection on what the program is entailing.

Resources to continue with "the rest of your life", next steps. Group sharing of global experiences with the program Brief closing practice

RETREAT DAY In addition to the 8 sessions, a small silent retreat is held on a Saturday, which is a day of intensive practice (approximately 8 hours). On this day consecutive practices are performed, including some different sitting meditation such as mountain meditation, loving-kindness or lake meditation.

ELIGIBILITY:
Inclusion Criteria:

* Working in a hospital
* Proficiency in the Spanish language

Exclusion Criteria:

* Have severe mental disorders.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2021-05-03 (Actual); Primary Completion 2021-10-10 (Actual); Study Completion 2021-10-10 (Actual)

PRIMARY OUTCOMES:
Symptoms Checklist 90 Revised (SCL-90-R) | Baseline, and 2 months
  This is a 90-item scale scored using a 5-point Likert scale from 0 (never) to 4 (extremely). This instrument is used to assess 9 dimensions: Somatization, Obsession-compulsion, Interpersonal sensitivity, Depression, Anxiety, Hostility, Phobic anxiety, Paranoid ideation, and Psychoticism. The scale also has 7 extra items distributed among 3 global indexes of distress: the GSI, which measures overall psychological distress; the PSDI, which is used to measure the intensity of symptoms; and Positive Symptom Total, used to measure the number of self-reported symptoms. Using the author´s instructions, the scores are transformed to percentiles (0-100). Percentiles ≥ 70 represent clinical symptoms in any of the subscale of this instrument.

SECONDARY OUTCOMES:
Perceived Stress Scale (PSS) | Baseline, and 2 months
  The PSS provides information on the perception of general stress during the preceding month. It consists on 14 items scores on a 5-point Likert scale (0 = never, 1 = almost never, 2 = once in a while, 3 = often, 4 = very often). Scores range from 0-56 (higher scores represent higher levels of stress)
Self-Compassion Scale (SCS) | Baseline, and 2 months
  The SCS is a 26-item self-reporting questionnaire with a 5-point Likert response format (from 1 = almost never to 5 = almost always).
Scale of Body Connection (SBC) | Baseline, and 2 months
  The SBC is a 20-item scale involving two distinct dimensions: Body Awareness and Bodily Dissociation. Rated on a 5-point Likert scale ranging from 1 (not at all) to 5 (all the time).
Five Facet Mindfulness Questionnaire (FFMQ) | Baseline, and 2 months
  The scale has 39 items and is answered with a 5-point Likert scale ranging from 1 (never) to 5 (always).

CONTACTS AND LOCATIONS:
Locations (1):
- Jose A. Puertas-Gonzalez, Granada, Spain